CLINICAL TRIAL: NCT03396042
Title: Natural History Study of CEP290-Related Retinal Degeneration
Status: Completed | Type: Observational
Sponsor: Editas Medicine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EDIT-NHS01
Record Dates: First submitted 2017-12-04; First posted 2018-01-10 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Blindness; Leber Congenital Amaurosis 10; Vision Disorders; Eye Diseases; Eye Diseases, Hereditary; Eye Disorders Congenital; Retinal Disease; Retinal Degeneration
Keywords: CEP290; LCA10; Retinal degenerative diseases (RDD); Leber congenital amaurosis (LCA); Congenital Retinal Blindness; p.Cys998X; c.2991+1655A>G; Eye Diseases Signs and Symptoms; Genetic Diseases, Inborn; Congenital Abnormalities; Eye Abnormalities
MeSH Terms: conditions — Blindness; Leber Congenital Amaurosis 10; Vision Disorders; Eye Diseases; Eye Diseases, Hereditary; Eye Abnormalities; Retinal Diseases; Retinal Degeneration; Meckel Syndrome, Type 4; Leber Congenital Amaurosis; Genetic Diseases, Inborn; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling for genetic testing of the CEP290 gene, including coding and intron 26 sequences, as part of a 280-gene retinal dystrophy gene panel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Group 1: 5 Patient target, ages 3 to 5 yr, with visual acuity Light Perception (LP) to <=20/200
- Group 2: 5 Patient target, ages 3 to 5 yr, with visual acuity >20/200 to <=20/50
- Group 3: 5 Patient target, ages 6 to 11 yr, with visual acuity LP to <=20/200
- Group 4: 5 Patient target, ages 6 to 11 yr, with visual acuity >20/200 to <=20/50
- Group 5: 5 Patient target, ages 12 to 17 yr, with visual acuity LP to <=20/200
- Group 6: 5 Patient target, ages 12 to 17 yr, with visual acuity >20/200 to <=20/50
- Group 7: 5 Patient target, ages 18yr and older, with visual acuity LP to <=20/200
- Group 8: 5 Patient target, ages 18yr and older, with visual acuity >20/200 to <=20/50

SUMMARY:
A prospective natural history study with systematic assessments and uniform follow-up to provide a high-quality dataset for assisting in the design of future clinical treatment trials involving patients with CEP290-related retinal degeneration caused by the common intron 26 mutation.

DETAILED DESCRIPTION:
The purpose of the study is to describe the natural history of CEP290-related retinal degeneration caused by a compound heterozygous or homozygous intron 26 c.2991+1655A>G mutation and to better understand the best assessments for evaluation of patients with this condition in a future interventional trial. Patients meeting the entry criteria will be enrolled in the study. Visits will occur at Screening, Baseline, and Months 3, 6, and 12, for a total duration of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient and/or parent/legal guardian must complete/sign an informed consent form (ICF). If required on a per patient basis, provisions can be made for alternative forms of consent (eg, witnessed consent). Where required by the IRB/IEC, minors must also verbalize or sign a confirmation of assent.
* At least 3 years of age at screening.
* Has abnormally decreased vision, defined as having light perception to 20/50 visual acuity in each eye, with examination and test results consistent with an inherited retinal degeneration due to mutations in the CEP290 gene.
* Has CEP290-related retinal degeneration caused by a compound heterozygous or homozygous intron 26 c.2991+1655A>G mutation (ie, 1 or 2 copies of the intron 26 c.2991+1655A>G mutation) confirmed by deoxyribonucleic acid sequencing.
* Has ability to cooperate with assessments relative to age.
* Has clear ocular media and adequate pupil dilation in at least 1 eye, to permit good quality fundus examination and optical coherence tomography (OCT) imaging.

Exclusion Criteria:

* Has history or current evidence of a medical condition (systemic or ophthalmic disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding) that may, in the opinion of the Investigator, preclude adherence to the scheduled study visits, safe participation in the study, or affect the results of the study (eg, uncontrolled systemic hypertension, autoimmune disease, advanced coronary artery disease, or cerebral vascular disease, other unstable or progressive cardiovascular, pulmonary, Parkinson's, liver or renal disease, cancer, or dementia).
* Has history or current evidence of ocular disease in either eye that, in the opinion of the Investigator, may confound assessment of this inherited retinal disease or the assessments utilized herein (eg, glaucoma, age-related macular degeneration, diabetic retinopathy, uveitis, or the presence of any condition that precludes adequate visualization of the fundus such as dense cataracts or corneal scarring).
* Achieves a passing score for the Visual Function Navigation Test at the maximum level of difficulty (ie, passes the most challenging Visual Function Navigation Test under the dimmest lighting conditions) with each eye independently and both eyes together.
* Is currently receiving gene therapy and/or has received gene therapy.
* Is currently enrolled in an investigational or interventional drug or device study and/or has participated in such a study within 30 days of Screening.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The indication for this study is CEP290-related retinal degeneration caused by a compound heterozygous or homozygous intron 26 c.2991+1655A>G mutation.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Characterize CEP290-related retinal degeneration | Through 12 months
  To prospectively characterize CEP290-related retinal degeneration and the clinical phenotype of patients with either compound heterozygous or homozygous intron 26 c.2991+1655A>G mutations

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Bascom Palmer Eye Institute, Miami, Florida
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - W.K. Kellogg Eye Center, Ann Arbor, Michigan
  - Casey Eye Institute - OHSU, Portland, Oregon
- Universite Pierre et Marie Curie, Paris, France
- Universitaetsklinikum Giessen and Marburg GmbH, Giessen, Germany
- Radboud Universitair Medisch Centrum, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No